CLINICAL TRIAL: NCT00940082
Title: The Cardiopathic Features and Analysis of Risk Factors in the Elderly Diabetic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Wu Qinan, Ethics Committee of Third Military Medical University, Third Military Medical University
Other Study IDs: the south west Hospital; Endocrine Department
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Two-Dimensional Echocardiography
Keywords: Diabetes;; Echocardiography;; High-sensitive C-reactive protein;; homocysteine;; TNF-α
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Take the fasting blood more than 12 hours overnight
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- youth control group: healthy people which ages from 30 to 59
- youth diabetes group: type 1 and type 2 diabetes patients which ages from 30 to 59
- the elderly diabetes group: type 1 and type 2 diabetes patients which ages from 60 to 90
- elderly control group: healthy people which ages from 60 to 90

SUMMARY:
Objectives: To investigate the cardiac condition of the diabetic patients in our hospital in order to seek for the new diagnostic method of warning its cardiovascular complications in early times.

Methods: 317 diabetic patients in our hospital from January in 2004 to July in 2008 were divided into 2 groups: group A (106 patients whose age ranged from (31-59) and group B (211 patients whose age ranged from (60-90). The height, weight, blood glucose, glycosylated hemoglobin, lipid, blood pressure, course of disease, ejection fraction (EF), fractional shortening(FS), diameter of left ventricle in late diastolic stage(LVEDd), the thickness of the ventricular septa（IVSDand the posterior wall of the right ventricle in late diastolic stage (LVPWd)were recorded respectively. Left ventricular mass index (LVMI), relative wall thickness (RWT) were calculated and High-sensitive C-reactive protein (HsCRP), homocysteine and TNF-α were detected. Multifactor logistic regression was made based on the comparison and contrast between all indexes to analyze the correlations between age and the positive indexes.

DETAILED DESCRIPTION:
Diabetes is one of the commonly seen health hazards in modern times. According to statistics, 70% people with diabetes have died of cardiovascular diseases.

Framingham 's study has proven the increase of the congestive heart-failure (2.4:1 in male patients and5:1 in female patients), which has no association with the age, hypertension, obesity, cardiovascular disease and Hyperlipidemia[1]. Other prospective studies also showed that the patients with diabetes in the early stage may be subject to abnormal echocardiogram and their probabilities of suffering from heart failure in the lifetime and Q-wave and non-Q wave myocardial infarction will be increased[1,2]. Early in 2000, American Heart Association issued a statement that "diabetes is a cardiovascular disease" [3]and in 2007, with reference to the joint guidelines concerning diabetes, pre-diabetes and cardiovascular disease, European Society of Cardiology (ESC) and the European Diabetes Research Institute (ESAD) clearly pointed out that hyperglycemia and cardiovascular disease (CVD) are closely related and the danger of CVD can be raised notably for those whose blood glucose is normal when fasting but tend to increase postprandially[4]. In the pathogenesis study of cardiovascular complications of diabetes, the promotion of oxidative stress and declination of the heart antioxidant reserves have close associations with the cardiovascular complications in animal and human body[5]. A number of cytokines and inflammatory signaling pathways are involved including tumor necrosis factor-α (TNF-α), high-sensitivity C-reactive protein (HsCRP), adiponectin, IL-6, NF-κB[1,6]. Accordingly, this study analyzes the echocardiography, high-sensitivity C-reactive protein and tumor necrosis factor-α of the patients with diabetics in our hospital in order to find early warning indicators of the cardiovascular complications of diabetes and provide prevention and treatment for cardiovascular complications of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* In-patient or out-patient patients diagnosed with diabetes
* Over 18 years of age
* Gender-open
* The type of diabetes (type 1 or type 2) open
* Patients receive a written informed consent to participate in the trial

Exclusion Criteria:

* those diabetic patients with acute and chronic infection, high blood pressure, special and Gestational diabetes Serious complications of heart, liver, lung, kidney damage Malignant tumors
* Pregnant women and breast-feeding women

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 1 and type 2 diabetic patients. They have been included in the standard diagnostic criteria for WHO1999 years and those diabetic patients with acute and chronic infection, high blood pressure, special and Gestational diabetic patients have been excluded. (Judgment have been made according to the case history, physical examination, medication, hormone history, blood routine etc) Those repeatedly hospitalized patients were recorded according to the time they took their first related inspection
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-06; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
the gender, height, weight, blood pressure, course of the disease of each patient was recorded | 1 day

SECONDARY OUTCOMES:
Left ventricular mass index (LVMI), relative wall thickness (RWT) were calculated and High-sensitive C-reactive protein (HsCRP), homocysteine and TNF-α were detected | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Chen Bing, doctor, Study Director — Endocrine Department, the south west Hospital of the Third Military Medical University
Locations (1):
- Endocrine Department, the First Affiliated Hospital of the Third Military Medical University, Chongqing, Chongqing Municipality, China